CLINICAL TRIAL: NCT03482011
Title: A Multicenter Study With a Randomized, Double-Blind, Placebo-Controlled Induction Dosing Period Followed by a Randomized Withdrawal Maintenance Dosing Period to Evaluate the Efficacy and Safety of Mirikizumab in Patients With Moderate-to-Severe Plaque Psoriasis OASIS-1
Brief Title: A Study to Evaluate the Efficacy and Safety of Mirikizumab (LY3074828) in Participants With Moderate-to-Severe Plaque Psoriasis
Acronym: OASIS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16505; I6T-MC-AMAK (Other: Eli Lilly and Company); 2017-003298-32 (EudraCT Number)
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-02-01

CONDITIONS: Psoriasis
Keywords: Psoriasis; IL-23
MeSH Terms: conditions — Psoriasis | interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirikizumab (Experimental): Induction Period:
  Participants received 250 milligrams (mg) mirikizumab administered subcutaneously (SC) every 4 weeks (Q4W).
  Maintenance Period:
  Participants received one of the four options below:
  Placebo administered SC every 8 weeks (Q8W) for responders (≥PASI 90).
  125 mg mirikizumab administered SC Q8W for responders (≥PASI 90).
  250 mg mirikizumab administered SC Q8W for responders (≥PASI 90).
  250 mg mirikizumab administered SC Q8W for non-responders (<PASI 90).
  Interventions: Drug: Mirikizumab
- Placebo (Placebo Comparator): Induction Period: Participants received placebo administered SC Q4W.
  Maintenance Period:
  Participants received one of the two options below:
  Placebo administered SC Q8W for responders (≥PASI 90).
  250 mg mirikizumab administered SC Q4W during week 16 to week 32 and Q8W during week 40 and 48 for non-responders (< PASI 90).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirikizumab — Administered SC
  Other Names: LY3074828
  Arms: Mirikizumab
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of mirikizumab in participants with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Present with chronic plaque psoriasis based on an investigator confirmed diagnosis of chronic psoriasis vulgaris for at least 6 months prior to baseline and meet the following criteria:

  * plaque psoriasis involving ≥10% BSA and absolute PASI score ≥12 in affected skin at screening and baseline
  * sPGA score of ≥3 at screening and baseline
* Candidate for systemic therapy and/or phototherapy for psoriasis.

Exclusion Criteria:

* Have an unstable or uncontrolled illness, including but not limited to a cerebro-cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurologic disease or abnormal laboratory values at screening, that in the opinion of the investigator, would potentially affect participant safety within the study or of interfering with the interpretation of data.
* Breastfeeding or nursing women.
* Have had serious, opportunistic, or chronic/recurring infection within 3 months prior to screening.
* Have received a Bacillus Calmette-Guerin (BCG) vaccination within 12 months or received live vaccine(s) (including attenuated live vaccines) within 12 weeks of baseline or intend to receive either during the study.
* Have any other skin conditions (excluding psoriasis) that would affect interpretation of the results.
* Have received systemic nonbiologic psoriasis therapy or phototherapy within 28 days prior to baseline.
* Have received topical psoriasis treatment within 14 days prior to baseline.
* Have received anti-tumor necrosis factor (TNF) biologics, or anti-interleukin (IL)-17 targeting biologics within 12 weeks prior to baseline.
* Have previous exposure to any biologic therapy targeting IL-23 (including ustekinumab), either licensed or investigational.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2020-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (69):
- United States (10):
  - Univ of Connecticut, Farmington, Connecticut
  - Florida Academic Dermatology Centers, Coral Gables, Florida
  - Renstar Medical Research, Ocala, Florida
  - Forward Clinical Trials, Inc, Tampa, Florida
  - Arlington Dermatology, Rolling Meadows, Illinois
  - The South Bend Clinic, South Bend, Indiana
  - Oregon Medical Research Center, Portland, Oregon
  - Dermatology and Skin Surgery Center, Exton, Pennsylvania
  - University of Utah MidValley Dematology, Murray, Utah
  - Multicare Health System, Tacoma, Washington
- Germany (7):
  - Gemeinschaftspraxis Mahlow, Mahlow, Brandenburg
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Praxis Gerlach, Dresden, Saxony
  - Charité Universitätsmedizin Berlin, Berlin
  - ISA GmbH, Berlin
  - Universitätsklinikum Hamburg - Eppendorf, Hamburg
  - Clinical Research Hamburg GmbH, Hamburg
- Japan (12):
  - Toho University School of Medicine, Sakura Hospital, Sakura, Chiba
  - Takagi Dermatological Clinic, Obihiro, Hokkaido
  - Kanto Rosai Hospital, Kawasaki, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Ryukyu University Hospital, Nakagami-gun, Okinawa
  - Kume Clinic, Nishi-ku Sakai-shi, Osaka
  - Shimane University Hospital, Izumo, Shimane
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-KU, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Seibo Hospital, Shinjuku-ku, Tokyo
  - Shirasaki Clinic, Takaoka-shi, Toyama
- Mexico (8):
  - Centro Medico del Angel S.C., Mexicali, Estado de Baja California
  - Instituto Dermatologico de Jalisco Dr. Jose Barba Rubio, Zapopan, Jalisco
  - Hospital de Jesus, Mexico City, Mexico City
  - Clínica Enfermedades Crónicas y Procedimientos Especiales SC, Morella, Michoacán
  - B&B Investigaciones Medicas, SC, Mazatlán, Sinaloa
  - Kohler Milstein Research, S.A. de C.V., Mérida, Yucatán
  - RM Pharma Specialists S.A. de C.V., Distrito Federal
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C, Durango
- Poland (5):
  - NZOZ ZDROWIE Osteo-Medic, Bialystok
  - "Dermed" Centrum Medyczne Sp. z o.o., Lodz
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - Centrum Medyczne AMED, Warsaw
  - DermMEDICA Sp. z o.o., Wroclaw
- Puerto Rico (2):
  - Office of Dr. Alma M. Cruz, Carolina, PR
  - GCM Medical Group PSC, San Juan, PR
- Russia (6):
  - GBUZ Clinical dermatology and venereological dispensary, Krasnodar
  - State scientific centre for dermatovenerology and cosmetolog, Moscow
  - First Moscow State Medical University n.a. Sechenov, Moscow
  - SPb SBHI Skin-venerologic dispensary #10, Saint Petersburg
  - GOU VPO 'Smolensk State Medical Academy of Ministry of Health and Social Development of Russian Federation', Smolensk
  - Tver State Medical University, Tver'
- South Korea (12):
  - Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Bundang CHA General Hospital, Sungnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Kyung Hee University Hospital, Seoul, Korea
  - Korea University Guro Hospital, Seoul, Korea
  - Ulsan University Hospital, Ulsan, Korea
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Severance Hospital Yonsei University Health System, Seoul
  - Hanyang University Medical Center, Seoul
  - Konkuk University Hospital, Seoul
- Taiwan (7):
  - National Taiwan University Hospital, Taipei, Zhongzheng District
  - National Taiwan University Hospital Hsin-Chu, Hsinchu
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - Taipei Medical University- Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital - Linkou, Taoyuan Hsien

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Hsieh CY, Hsu FL, Tsai TF. Comparison of Drug-Free Remission after the End of Phase III Trials of Three Different Anti-IL-23 Inhibitors in Psoriasis. Dermatol Ther (Heidelb). 2024 Sep;14(9):2607-2620. doi: 10.1007/s13555-024-01229-6. Epub 2024 Jul 29. PMID 39073712

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Q4W: Induction Period: Participants received placebo administered subcutaneously (SC) every 4 weeks (Q4W).
- 250 mg Miri Q4W: Induction Period: Participants received 250 milligrams (mg) mirikizumab (miri) administered SC Q4W.
- Placebo Q4W to Placebo Q8W (Placebo Responder): Maintenance Period: Participants received placebo administered SC every 8 weeks (Q8W). Responders had ≥PASI 90.
  Participants had received placebo administered SC Q4W during induction period.
  Follow-up Period: Participants did not receive drug during the follow-up period.
- Placebo Q4W to 250 mg Miri Q4W /Q8W (Placebo Non-Responders): Maintenance Period: Participants received 250 mg mirikizumab administered SC Q4W during week 16 to week 32 and Q8W during week 40 and 48. Non-responders had < PASI 90.
  Participants had received placebo administered SC Q4W during induction period.
  Follow-up Period: Participants did not receive drug during the follow-up period.
- 250 mg Miri Q4W Responders to Placebo Q8W: Maintenance Period: Participants received placebo administered SC Q8W. Responders had ≥PASI 90.
  Participants had received 250 mirikizumab administered SC Q4W during induction period.
  Follow-up Period: Participants did not receive drug during the follow-up period.
- 250 mg Miri Q4W Responders to 125 mg Miri Q8W: Maintenance Period: Participants received 125 mg mirikizumab administered SC Q8W. Responders had ≥PASI 90.
  Participants had received 250 mirikizumab administered SC Q4W during induction period.
  Follow-up Period: Participants did not receive drug during the follow-up period.
- 250 mg Miri Q4W Responder to 250 mg Miri Q8W: Maintenance Period: Participants received 250 mg mirikizumab administered SC Q8W. Responders had ≥PASI 90.
  Participants had received 250 mirikizumab administered SC Q4W during induction period.
  Follow-up Period: Participants did not receive drug during the follow-up period.
- 250 mg Miri Q4W to 250 mg Miri Q8W (Miri Non-Responders): Maintenance Period: Participants received 250 mg mirikizumab administered SC Q8W. Non-responders had < PASI 90.
  Participants had received 250 mirikizumab administered SC Q4W during induction period.
  Follow-up Period: Participants did not receive drug during the follow-up period.
Period: Induction Period (16 Weeks)
Arm/Group | Placebo Q4W | 250 mg Miri Q4W | Placebo Q4W to Placebo Q8W (Placebo Responder) | Placebo Q4W to 250 mg Miri Q4W /Q8W (Placebo Non-Responders) | 250 mg Miri Q4W Responders to Placebo Q8W | 250 mg Miri Q4W Responders to 125 mg Miri Q8W | 250 mg Miri Q4W Responder to 250 mg Miri Q8W | 250 mg Miri Q4W to 250 mg Miri Q8W (Miri Non-Responders)
Started | 107 | 423 | 0 (Participants were assigned to this arm during maintenance period.) | 0 (Participants were assigned to this arm during maintenance period.) | 0 (Participants were assigned to this arm during maintenance period.) | 0 (Participants were assigned to this arm during maintenance period.) | 0 (Participants were assigned to this arm during maintenance period.) | 0 (Participants were assigned to this arm during maintenance period.)
Received at Least One Dose of Study Drug | 107 | 422 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 101 | 412 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Screen Failure | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period (36 Weeks)
Arm/Group | Placebo Q4W | 250 mg Miri Q4W | Placebo Q4W to Placebo Q8W (Placebo Responder) | Placebo Q4W to 250 mg Miri Q4W /Q8W (Placebo Non-Responders) | 250 mg Miri Q4W Responders to Placebo Q8W | 250 mg Miri Q4W Responders to 125 mg Miri Q8W | 250 mg Miri Q4W Responder to 250 mg Miri Q8W | 250 mg Miri Q4W to 250 mg Miri Q8W (Miri Non-Responders)
Started | 0 (Participants were assigned to this arm during induction period.) | 0 (Participants were assigned to this arm during induction period.) | 7 | 94 | 91 | 90 | 91 | 140
Relapse | 0 | 0 | 1 | 0 | 41 | 3 | 2 | 0
Roll Over to I6T-MC-AMAH (NCT03556202) | 0 | 0 | 6 | 88 | 86 | 85 | 87 | 121
Completed | 0 | 0 | 6 | 90 | 86 | 86 | 87 | 123
Not Completed | 0 | 0 | 1 | 4 | 5 | 4 | 4 | 17
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 2
Period: Follow-up Period (12 Weeks)
Arm/Group | Placebo Q4W | 250 mg Miri Q4W | Placebo Q4W to Placebo Q8W (Placebo Responder) | Placebo Q4W to 250 mg Miri Q4W /Q8W (Placebo Non-Responders) | 250 mg Miri Q4W Responders to Placebo Q8W | 250 mg Miri Q4W Responders to 125 mg Miri Q8W | 250 mg Miri Q4W Responder to 250 mg Miri Q8W | 250 mg Miri Q4W to 250 mg Miri Q8W (Miri Non-Responders)
Started | 0 (Participants were assigned to this arm during induction period.) | 0 (Participants were assigned to this arm during induction period.) | 1 | 10 | 2 | 4 | 4 | 21
Completed | 0 | 0 | 0 | 5 | 2 | 3 | 2 | 4
Not Completed | 0 | 0 | 1 | 5 | 0 | 1 | 2 | 17
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 6
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 250 mg Miri Q4W: Induction Period: Participants received 250 mg mirikizumab administered SC Q4W.
- Total: Total of all reporting groups
Arm/Group | Placebo Q4W | 250 mg Miri Q4W | Total
Number analyzed (Participants) | 107 | 423 | 530
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (13.70) | 46.4 (13.56) | 46.3 (13.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 124 | 157
  Male | 74 | 299 | 373
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 13 | 17
  Not Hispanic or Latino | 11 | 53 | 64
  Unknown or Not Reported | 92 | 357 | 449
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 50 | 64
  Asian | 33 | 139 | 172
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 2 | 6
  White | 56 | 231 | 287
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 11 | 45 | 56
  Puerto Rico | 5 | 15 | 20
  United States | 16 | 69 | 85
  Japan | 10 | 44 | 54
  Taiwan | 12 | 49 | 61
  Poland | 11 | 44 | 55
  Mexico | 15 | 61 | 76
  Germany | 16 | 58 | 74
  Russia | 11 | 38 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Static Physician's Global Assessment of (sPGA) (0,1) With at Least a 2-point Improvement From Baseline
Description: The sPGA is the physician's determination of the participant's psoriasis (PsO) lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participant's PsO was assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a post-baseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline.
Time Frame: Week 16
Population: Induction Period: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 107 | 423
Percentage of participants | 6.5 [1.9 to 11.2] | 69.3 [64.9 to 73.7]
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 63.0, 95% CI 2-sided [56.5 to 69.4]

2. Primary Outcome: Percentage of Participants Achieving a ≥90% Improvement From Baseline in Psoriasis Area and Severity Score (PASI 90)
Description: PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of scaling, redness, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis (PsO) to 72 for the most severe disease. For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no PsO) to 72 (the most severe disease).
Time Frame: Week 16
Population: Induction Period: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 107 | 423
Percentage of participants | 6.5 [1.9 to 11.2] | 64.3 [59.7 to 68.9]
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 57.8, 95% CI 2-sided [51.3 to 64.4]

3. Secondary Outcome: Percentage of Participants Achieving a ≥75% Improvement From Baseline in PASI (PASI 75)
Description: as for outcome 2
Time Frame: Week 4
Population: Induction Period: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 107 | 423
Percentage of participants | 0.9 [0.0 to 2.8] | 17.0 [13.4 to 20.6]
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.6, 95% CI 2-sided [11.6 to 19.7]

4. Secondary Outcome: Percentage of Participants Achieving a ≥75% Improvement From Baseline in PASI (PASI 75)
Description: as for outcome 2
Time Frame: Week 16
Population: Induction Period: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 107 | 423
Percentage of participants | 9.3 [3.8 to 14.9] | 82.5 [78.9 to 86.1]
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 73.6, 95% CI 2-sided [67.1 to 80.1]

5. Secondary Outcome: Percentage of Participants Achieving a ≥100% Improvement From Baseline in Psoriasis Area and Severity Score (PASI 100)
Description: as for outcome 2
Time Frame: Week 16
Population: Induction Period: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 107 | 423
Percentage of participants | 0.9 [0.0 to 2.8] | 32.4 [27.9 to 36.8]
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 30.8, 95% CI 2-sided [26.0 to 35.7]

6. Secondary Outcome: Percentage of Participants With ≤1% of Body Surface Area (BSA) With Psoriasis Involvement
Description: The BSA is the percentage involvement of psoriasis on each participant's body surface on a continuous scale from 0% (no involvement) to 100% (full involvement), in which 1% corresponds to the size of the participant's hand (including the palm, fingers, and thumb). The total BSA affected was the summation of individual regions affected. Percentage response is calculated by number of participants with a response divided by number of participants with non-missing values multiplied by 100.
Time Frame: Week 16
Population: Induction Period:All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 107 | 423
Percentage of participants | 0.9 [0.0 to 2.8] | 49.2 [44.4 to 53.9]
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 48.1, 95% CI 2-sided [42.9 to 53.2]

7. Secondary Outcome: Percentage of Participants With a Psoriasis Symptoms Scale (PSS) Symptoms Score of 0 in Those With a PSS Symptoms Score ≥1 at Baseline
Description: PSS is a patient-administered assessment of 4 symptoms (itch, pain, stinging, and burning); 3 signs (redness, scaling, and cracking); and 1 item on the discomfort related to symptoms/signs. The overall severity for each individual symptom/sign from the patient's psoriasis is indicated by selecting the number from a numeric rating scale (NRS) of 0 to 10 that best describes the worst level of each symptom/sign in the past 24 hours, where 0=no symptom/sign and 10=worst imaginable symptom/sign. In addition, a symptoms score ranging from 0 (no symptoms) to 40 (worst imaginable symptoms), and a signs score of 0 (no signs) to 30 (worst imaginable signs) will be reported. Percentage response is calculated by number of participants with a response divided by number of participants with non-missing values multiplied by 100.
Time Frame: Week 16
Population: Induction Period: All randomized participants who had PSS symptoms score ≥1 at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 105 | 410
percentage of participants | 0 [0.0 to 0.0] | 19.0 [15.2 to 22.8]
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 18.3, 95% CI 2-sided [14.5 to 22.1]

8. Secondary Outcome: Percentage of Participants Achieving a Dermatology Life Quality Index (DLQI) Total Score of (0,1) With at Least a 5-Point Improvement (Reduction) From Baseline in Participants With a Baseline DLQI Total Score ≥5
Description: The DLQI is a patient-reported, 10-question, quality-of-life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". For all questions, if unanswered the question is scored as "0". Totals range from 0 to 30 (less to more impairment). A DLQI total score of 0 to 1 is considered as having no effect on a patient's health-related quality of life (HRQoL), and a 5-point change from baseline is considered as the minimal clinically important difference (MCID) threshold. Percentage response is calculated by number of participants with a response divided by number of participants with non-missing values multiplied by 100.
Time Frame: Week 16
Population: Induction Period: All randomized participants who had a baseline DLQI Total Score ≥5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 92 | 384
Percentage of participants | 5.4 [0.8 to 10.1] | 54.7 [49.7 to 59.7]
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 49.6, 95% CI 2-sided [42.8 to 56.4]

9. Secondary Outcome: Percentage of Participants Maintaining Clinical Response (PASI 90) After Re-randomization at the Start of the Randomized Withdrawal Period
Description: as for outcome 2
Time Frame: Week 52
Population: Maintenance Period: All re-randomized participants who were responders (≥PASI 90).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 250 mg Miri Q4W Responders to Placebo Q8W: Maintenance Period: Participants received placebo administered SC Q8W. Responders had ≥PASI 90.
  Participants had received 250 mirikizumab administered SC Q4W during induction period.
- 250 mg Miri Q4W Responders to 125 mg Miri Q8W: Maintenance Period: Participants received 125 mg mirikizumab administered SC Q8W. Responders had ≥PASI 90.
  Participants had received 250 mirikizumab administered SC Q4W during induction period.
- 250 mg Miri Q4W Responder to 250 mg Miri Q8W: Maintenance Period: Participants received 250 mg mirikizumab administered SC Q8W. Responders had ≥PASI 90.
  Participants had received 250 mirikizumab administered SC Q4W during induction period.
Arm/Group | 250 mg Miri Q4W Responders to Placebo Q8W | 250 mg Miri Q4W Responders to 125 mg Miri Q8W | 250 mg Miri Q4W Responder to 250 mg Miri Q8W
Number analyzed (Participants) | 91 | 90 | 91
Percentage of participants | 18.7 [10.7 to 26.7] | 85.6 [78.3 to 92.8] | 84.6 [77.2 to 92.0]
Statistical Analysis 1: Comparison: 250 mg Miri Q4W Responders to Placebo Q8W vs 250 mg Miri Q4W Responders to 125 mg Miri Q8W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 66.7, 95% CI 2-sided [56.0 to 77.5]
Statistical Analysis 2: Comparison: 250 mg Miri Q4W Responders to Placebo Q8W vs 250 mg Miri Q4W Responder to 250 mg Miri Q8W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 65.9, 95% CI 2-sided [54.9 to 77.0]

10. Secondary Outcome: Change in Palmoplantar Psoriasis Severity Index (PPASI) Total Score in Participants With Palmoplantar Involvement at Baseline
Description: The Palmoplantar PASI is a composite score derived from the sum scores for erythema, induration, and desquamation multiplied by a score for the extent of palm and sole area involvement, ranging from 0 (no PPASI) to 72 (most severe PPASI). The PPASI was only assessed if participants have palmoplantar psoriasis at baseline. Least Squares Mean (LS Mean) was calculated using mixed model repeated measures (MMRM) model with treatment, baseline value, visit, the interaction of the baseline value-by-visit, the interaction of treatment by-visit, and previous exposure to biologic therapy (yes/no), body weight (<100 kg or >=100 kg), and geographic region (North America or Other) as covariates.
Time Frame: Week 16
Population: Induction Period: All randomized participants who had palmoplantar involvement at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 24 | 111
score on a scale | -1.13 (1.29) | -5.83 (0.72)
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -4.70, 95% CI 2-sided [-7.31 to -2.10], Standard Error of Mean 1.32

11. Secondary Outcome: Change in Psoriasis Scalp Severity Index (PSSI) Total Score in Participants With Scalp Involvement at Baseline
Description: The PSSI is a physician assessment of erythema, induration and desquamation and percent of scalp that is covered with a scores range from 0 (none) to 4 (very severe). The composite score is derived from the sum of scores for erythema, induration, and desquamation multiplied by the score recorded for the extent of the scalp area involved, 1 (<10%) to 6 (90%-100%) with a total score ranging from 0 (less severity) to 72 (more severity). LS Mean was calculated using MMRM model with treatment, baseline value, visit, the interaction of the baseline value-by-visit, the interaction of treatment by-visit, and previous exposure to biologic therapy (yes/no), body weight (<100 kg or >=100 kg), and geographic region (North America or Other) as covariates.
Time Frame: Week 16
Population: Induction Period: All randomized participants who had scalp Involvement at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 94 | 381
score on a scale | -2.70 (0.95) | -20.03 (0.55)
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -17.33, 95% CI 2-sided [-19.28 to -15.39], Standard Error of Mean 0.99

12. Secondary Outcome: Change in Nail Psoriasis Severity Index (NAPSI) Total Score in Participants With Fingernail Involvement at Baseline
Description: The NAPSI scale is used to evaluate the severity of fingernail bed Ps and fingernail matrix PsO by area of involvement. The fingernail is divided into quadrants. Each fingernail is given a score for fingernail bed PsO 0 (none) to 4 (PsO in 4 quadrants of the fingernail) and fingernail matrix PsO 0 (none) to 4 (Ps in 4 quadrants of the matrix), depending on the presence (score of 1) or absence (score of 0) of any of the features of fingernail bed or matrix PsO in each quadrant. The sum of all fingernails equals the total NAPSI score range is from 0 (no effect) to 80 (more severe psoriasis). LS Mean was calculated using MMRM model with treatment, baseline value, visit, the interaction of the baseline value-by-visit, the interaction of treatment by-visit, and previous exposure to biologic therapy (yes/no), body weight (<100 kg or >=100 kg), and geographic region (North America or Other) as covariates.
Time Frame: Week 16
Population: Induction Period: All randomized participants who had Nail Psoriasis involvement at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 64 | 248
score on a scale | -2.04 (1.60) | -9.01 (0.89)
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -6.98, 95% CI 2-sided [-10.37 to -3.58], Standard Error of Mean 1.73

13. Secondary Outcome: Change From Baseline on the Short Form (SF)-36 Physical Component Summary (PCS)
Description: SF-36 consists of 36 questions measuring 8 health domains: physical functioning, bodily pain, role limitations due to physical problems, role limitations due to emotional problems, general health perceptions, mental health, social function, and vitality. The patient's responses are solicited using Likert scales that vary in length, with 3-6 response options per item. The SF-36 can be scored into the 8 health domains named above and two overall summary scores: physical component summary (PCS) and mental component summary (MCS) scores. The domain and summary scores range from 0 to 100; higher scores indicate better levels of function and/or better health. LS Mean was calculated using Analysis of covariance (ANCOVA) model with treatment and baseline value, previous exposure to biologic therapy (yes/no), body weight (<100 kg or >=100 kg), and geographic region (North America or Other) as fixed factors.
Time Frame: Baseline, Week 16
Population: Induction Period: All randomized participants who had a baseline and at least one post-baseline PCS value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 106 | 418
score on a scale | 0.35 (0.69) | 5.21 (0.43)
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 4.86, 95% CI 2-sided [3.50 to 6.22], Standard Error of Mean 0.69

14. Secondary Outcome: Change From Baseline on the SF-36 Mental Component Summary (MCS)
Description: as for outcome 13
Time Frame: Baseline, Week 16
Population: Induction Period: All randomized participants who had a baseline and at least one post-baseline MCS value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 106 | 418
score on a scale | 0.32 (0.73) | 5.10 (0.46)
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 4.78, 95% CI 2-sided [3.33 to 6.23], Standard Error of Mean 0.74

15. Secondary Outcome: Percentage of Participants With Patient's Global Assessment of Psoriasis (PatGA (0,1)) and >=2 Improvement From Baseline
Description: The PatGA is a single-item self-reported instrument asking the participant to rate the severity of their psoriasis "today" by circling a number on the numeric rating scale from 0 (Clear = no psoriasis) to 5 (Severe = the worst their psoriasis has ever been). Percentage response is calculated by number of participants with a response divided by number of participants with non-missing values multiplied by 100.
Time Frame: Baseline, Week 16
Population: Induction Period: All randomized participants who had a baseline >= 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 104 | 419
Percentage of participants | 1.0 [0.0 to 2.8] | 69.5 [65.0 to 73.9]
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 68.1, 95% CI 2-sided [63.2 to 72.9]

16. Secondary Outcome: Change From Baseline on the Work Productivity and Activity Impairment Questionnaire: Psoriasis (WPAI-PSO)
Description: The WPAI-PSO consists of 6 questions to determine employment status, hours missed from work because of psoriasis, hours missed from work for other reasons, hours actually worked, the degree to which psoriasis affected work productivity while at work, and the degree to which psoriasis affected activities outside of work. Four scores are derived: absenteeism, presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism and impairment in activities performed outside of work. Each WPAI score is expressed as impairment percentages (0-100) with higher numbers indicating greater impairment and less productivity, that is, worse outcomes. LS Mean was calculated using Analysis of covariance (ANCOVA) model with treatment and baseline value, previous exposure to biologic therapy (yes/no), body weight (<100 kg or >=100 kg), and geographic region (North America or Other) as fixed factors.
Time Frame: Baseline, Week 16
Population: Induction Period:All randomized participants who had a baseline and at least one post-baseline WPAI-PSO value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 106 | 418
score on a scale
  Absenteeism: number analyzed (Participants) | 65 | 277
  Absenteeism | 0.10 (1.87) | -3.57 (1.12)
  Presenteeism: number analyzed (Participants) | 64 | 271
  Presenteeism | -4.54 (2.39) | -24.79 (1.42)
  Overall Absenteeism and Presenteeism: number analyzed (Participants) | 64 | 271
  Overall Absenteeism and Presenteeism | -3.45 (2.82) | -24.54 (1.68)
  Impairment in Activities Performed Outside of Work | -6.83 (2.27) | -29.73 (1.41)
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Absenteeism; Test type: Superiority; p = 0.002, ANOVA; Mean Difference (Net) = -3.68, 95% CI 2-sided [-7.30 to -0.06], Standard Error of Mean 1.84
Statistical Analysis 2: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Presenteeism; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -20.24, 95% CI 2-sided [-24.89 to -15.60], Standard Error of Mean 2.37
Statistical Analysis 3: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Overall Absenteeism and Presenteeism; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -21.09, 95% CI 2-sided [-26.56 to -15.62], Standard Error of Mean 2.78
Statistical Analysis 4: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Impairment in Activities Performed Outside of Work; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -22.91, 95% CI 2-sided [-27.39 to -18.43], Standard Error of Mean 2.28

17. Secondary Outcome: Change From Baseline in Quick Inventory of Depressive Symptomology (QIDS-SR16) Total Score in Those With a Baseline QIDS-SR16 Total Score ≥11
Description: QIDS-SR16 is a participant-administered, 16-item instrument intended to assess the existence and severity of symptoms of depression. A participant is asked to consider each statement as it relates to the way they have felt for the past 7 days and rate each on a 4-point scale: 0 (best) to 3 (worst). The sum of the 16 items corresponding to 9 depression domains [sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance (initial, middle and late insomnia or hypersomnia), decrease/increase in appetite/weight, and psychomotor agitation/retardation] to give a single total scores range from 0 to 27, with higher scores indicating greater symptom severity. Whereas 0-5 indicates no symptoms. LS Mean was calculated using ANCOVA model with treatment and baseline value, previous exposure to biologic therapy (yes/no), body weight (<100 kg or >=100 kg), and geographic region (North America or Other) as fixed factors.
Time Frame: Baseline, Week 16
Population: Induction Period: All participants who received at least one dose of study drug who had a baseline QIDS-SR16 total score >=11.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 10 | 35
score on a scale | -4.95 (1.94) | -4.42 (1.43)
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p = 0.004, ANCOVA; Mean Difference (Net) = 0.53, 95% CI 2-sided [-3.08 to 4.14], Standard Error of Mean 1.79

18. Secondary Outcome: Percentage of Participants Achieving a Dermatology Life Quality Index (DLQI) (0,1)
Description: as for outcome 8
Time Frame: Week 16
Population: Induction Period: All randomized participants who had a baseline and at least one post-baseline DLQI value.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Q4W | 250 mg Miri Q4W
Number analyzed (Participants) | 104 | 413
Percentage of participants | 8.7 [3.3 to 14.1] | 57.1 [52.4 to 61.9]
Statistical Analysis 1: Comparison: Placebo Q4W vs 250 mg Miri Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 48.8, 95% CI 2-sided [41.6 to 55.9]

19. Secondary Outcome: Induction Period: Pharmacokinetics (PK): Minimum Observed Serum Concentration at Steady State (Ctrough,ss) of Mirikizumab at Week 16
Description: Minimum observed serum concentration at steady state (Ctrough,ss) of mirikizumab at Week 16.
Time Frame: Week 16: Day 113
Population: Induction Period: All participants who received at least one dose of study drug who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter(micrograms/mL)
Arm/Group | 250 mg Miri Q4W
Number analyzed (Participants) | 387
micrograms per milliliter(micrograms/mL) | 2.00 (139)

ADVERSE EVENTS:
Time Frame: Baseline Up To 64 Weeks
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- 250 mg Miri Q4W: Induction Period: Participants received 250 mg mirikizumab (miri) administered SC Q4W.
- Placebo Q4W to Placebo Q8W (Placebo Responder): Maintenance Period: Participants received placebo administered SC Q8W. Responders had ≥PASI 90.
  Participants had received placebo administered SC Q4W during induction period.
- Placebo Q4W to 250 mg Miri Q4W /Q8W (Placebo Non-Responders): Maintenance Period: Participants received 250 mg mirikizumab administered SC Q4W during week 16 to week 32 and Q8W during week 40 and 48. Non-responders had < PASI 90.
  Participants had received placebo administered SC Q4W during induction period.
- 250mg Miri Q4W to 250mg Miri Q8W(Miri Non-Responders): Maintenance Period: Participants received 250 mg mirikizumab administered SC Q8W. Non-responders had < PASI 90.
  Participants had received 250 mirikizumab administered SC Q4W during induction period.
- Relapse: Participants that relapsed were in the following arms:
  Placebo Q4W to Placebo Q8W (Placebo Responder).
  250 mg Miri Q4W Responders to Placebo Q8W.
  250 mg Miri Q4W Responders to 125 mg Miri Q8W.
  250 mg Miri Q4W Responder to 250 mg Miri Q8W.
- Placebo Q4W to Placebo Q8W (Responder) Follow-up Period; Placebo Q4W to Placebo Non-Responder-Follow-up Period; 250 mg Miri Q4W to Placebo Q8W (Responders) Follow-up Period; 250mg Miri Q4W to 125 mg Miri Q8W(Responders) Follow-up Period; 250mg Miri Q4W to 250mg Miri Q8W(Responders) Follow-up Period; 250 Miri Q4W to Miri Nonresponder-Follow-up Period: Follow-up Period: Participants did not receive drug during the follow-up period.
- Placebo Q4W Discontinued During Induction-Follow-up Period: Follow-up Period: Participants did not receive drug during the follow-up period.
  Participants discontinued (DC) before induction week 16 and counted as placebo non-responders.
- 250 Miri Q4W Discontinued During Induction-Follow-up: Follow-up Period: Participants did not receive drug during the follow-up period.
  Participants discontinued (DC) before induction week 16 and counted as miri non-responders.
Arm/Group | Placebo Q4W | 250 mg Miri Q4W | Placebo Q4W to Placebo Q8W (Placebo Responder) | Placebo Q4W to 250 mg Miri Q4W /Q8W (Placebo Non-Responders) | 250 mg Miri Q4W Responders to Placebo Q8W | 250 mg Miri Q4W Responders to 125 mg Miri Q8W | 250 mg Miri Q4W Responder to 250 mg Miri Q8W | 250mg Miri Q4W to 250mg Miri Q8W(Miri Non-Responders) | Relapse | Placebo Q4W to Placebo Q8W (Responder) Follow-up Period | Placebo Q4W Discontinued During Induction-Follow-up Period | Placebo Q4W to Placebo Non-Responder-Follow-up Period | 250 mg Miri Q4W to Placebo Q8W (Responders) Follow-up Period | 250mg Miri Q4W to 125 mg Miri Q8W(Responders) Follow-up Period | 250mg Miri Q4W to 250mg Miri Q8W(Responders) Follow-up Period | 250 Miri Q4W Discontinued During Induction-Follow-up | 250 Miri Q4W to Miri Nonresponder-Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/422 | 0/7 | 0/94 | 0/91 | 0/90 | 0/91 | 0/140 | 0/47 | 0/1 | 0/4 | 0/6 | 0/2 | 0/4 | 0/4 | 0/5 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/107 | 5/422 | 0/7 | 0/94 | 3/91 | 1/90 | 3/91 | 0/140 | 0/47 | 0/1 | 0/4 | 0/6 | 0/2 | 0/4 | 0/4 | 0/5 | 0/16
Other Adverse Events (participants affected / at risk) | 51/107 | 199/422 | 0/7 | 0/94 | 49/91 | 61/90 | 55/91 | 0/140 | 17/47 | 0/1 | 0/4 | 0/6 | 0/2 | 0/4 | 0/4 | 0/5 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q4W (N=107) | 250 mg Miri Q4W (N=422) | Placebo Q4W to Placebo Q8W (Placebo Responder) (N=7) | Placebo Q4W to 250 mg Miri Q4W /Q8W (Placebo Non-Responders) (N=94) | 250 mg Miri Q4W Responders to Placebo Q8W (N=91) | 250 mg Miri Q4W Responders to 125 mg Miri Q8W (N=90) | 250 mg Miri Q4W Responder to 250 mg Miri Q8W (N=91) | 250mg Miri Q4W to 250mg Miri Q8W(Miri Non-Responders) (N=140) | Relapse (N=47) | Placebo Q4W to Placebo Q8W (Responder) Follow-up Period (N=1) | Placebo Q4W Discontinued During Induction-Follow-up Period (N=4) | Placebo Q4W to Placebo Non-Responder-Follow-up Period (N=6) | 250 mg Miri Q4W to Placebo Q8W (Responders) Follow-up Period (N=2) | 250mg Miri Q4W to 125 mg Miri Q8W(Responders) Follow-up Period (N=4) | 250mg Miri Q4W to 250mg Miri Q8W(Responders) Follow-up Period (N=4) | 250 Miri Q4W Discontinued During Induction-Follow-up (N=5) | 250 Miri Q4W to Miri Nonresponder-Follow-up Period (N=16)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Q4W (N=107) | 250 mg Miri Q4W (N=422) | Placebo Q4W to Placebo Q8W (Placebo Responder) (N=7) | Placebo Q4W to 250 mg Miri Q4W /Q8W (Placebo Non-Responders) (N=94) | 250 mg Miri Q4W Responders to Placebo Q8W (N=91) | 250 mg Miri Q4W Responders to 125 mg Miri Q8W (N=90) | 250 mg Miri Q4W Responder to 250 mg Miri Q8W (N=91) | 250mg Miri Q4W to 250mg Miri Q8W(Miri Non-Responders) (N=140) | Relapse (N=47) | Placebo Q4W to Placebo Q8W (Responder) Follow-up Period (N=1) | Placebo Q4W Discontinued During Induction-Follow-up Period (N=4) | Placebo Q4W to Placebo Non-Responder-Follow-up Period (N=6) | 250 mg Miri Q4W to Placebo Q8W (Responders) Follow-up Period (N=2) | 250mg Miri Q4W to 125 mg Miri Q8W(Responders) Follow-up Period (N=4) | 250mg Miri Q4W to 250mg Miri Q8W(Responders) Follow-up Period (N=4) | 250 Miri Q4W Discontinued During Induction-Follow-up (N=5) | 250 Miri Q4W to Miri Nonresponder-Follow-up Period (N=16)
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract subcapsular (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Defaecation disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival atrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (6) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fat necrosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 5 (20) | 22 (109) | 0 (0) | 0 (0) | 2 (48) | 5 (49) | 6 (65) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 5 (11) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Borrelia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0/74 (0) | 1/298 (1) | 0/3 (0) | 0/67 (0) | 0/61 (0) | 0/64 (0) | 0/59 (0) | 0/106 (0) | 0/31 (0) | 0 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0/2 (0) | 0/4 (0) | 0/9 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema migrans (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis a (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis e (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 14 (14) | 55 (61) | 0 (0) | 0 (0) | 15 (35) | 13 (16) | 9 (13) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0/33 (0) | 0/124 (0) | 0/4 (0) | 0/27 (0) | 0/30 (0) | 1/26 (1) | 0/32 (0) | 0/34 (0) | 0/16 (0) | 0 (0) | 0/1 (0) | 0 (0) | 0 (0) | 0 (0) | 0/2 (0) | 0/1 (0) | 0/7 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salpingo-oophoritis (Infections and infestations) | 0/33 (0) | 0/124 (0) | 0/4 (0) | 0/27 (0) | 0/30 (0) | 0/26 (0) | 1/32 (1) | 0/34 (0) | 0/16 (0) | 0 (0) | 0/1 (0) | 0 (0) | 0 (0) | 0 (0) | 0/2 (0) | 0/1 (0) | 0/7 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 16 (20) | 0 (0) | 0 (0) | 7 (17) | 5 (5) | 10 (11) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 8 (10) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0/33 (0) | 1/124 (1) | 0/4 (0) | 0/27 (0) | 0/30 (0) | 0/26 (0) | 0/32 (0) | 0/34 (0) | 1/16 (1) | 0 (0) | 0/1 (0) | 0 (0) | 0 (0) | 0 (0) | 0/2 (0) | 0/1 (0) | 0/7 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/33 (0) | 1/124 (1) | 0/4 (0) | 0/27 (0) | 0/30 (0) | 0/26 (0) | 0/32 (0) | 0/34 (0) | 0/16 (0) | 0 (0) | 0/1 (0) | 0 (0) | 0 (0) | 0 (0) | 0/2 (0) | 0/1 (0) | 0/7 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin d dimer increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis b dna assay positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroxine free decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Very low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiometabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overweight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (11) | 0 (0) | 0 (0) | 5 (12) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 3 (6) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 10 (10) | 0 (0) | 0 (0) | 2 (6) | 5 (9) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tobacco abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0/33 (0) | 0/124 (0) | 0/4 (0) | 0/27 (0) | 1/30 (2) | 0/26 (0) | 0/32 (0) | 0/34 (0) | 0/16 (0) | 0 (0) | 0/1 (0) | 0 (0) | 0 (0) | 0 (0) | 0/2 (0) | 0/1 (0) | 0/7 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/33 (0) | 0/124 (0) | 0/4 (0) | 0/27 (0) | 0/30 (0) | 1/26 (1) | 1/32 (2) | 0/34 (0) | 0/16 (0) | 0 (0) | 0/1 (0) | 0 (0) | 0 (0) | 0 (0) | 0/2 (0) | 0/1 (0) | 0/7 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/74 (0) | 0/298 (0) | 0/3 (0) | 0/67 (0) | 0/61 (0) | 0/64 (0) | 1/59 (1) | 0/106 (0) | 0/31 (0) | 0 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0/2 (0) | 0/4 (0) | 0/9 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0/33 (0) | 0/124 (0) | 0/4 (0) | 0/27 (0) | 1/30 (2) | 0/26 (0) | 0/32 (0) | 0/34 (0) | 0/16 (0) | 0 (0) | 0/1 (0) | 0 (0) | 0 (0) | 0 (0) | 0/2 (0) | 0/1 (0) | 0/7 (0)
Prostatitis (Reproductive system and breast disorders) | 0/74 (0) | 1/298 (1) | 0/3 (0) | 0/67 (0) | 0/61 (0) | 0/64 (0) | 0/59 (0) | 0/106 (0) | 0/31 (0) | 0 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0/2 (0) | 0/4 (0) | 0/9 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0/33 (0) | 1/124 (1) | 0/4 (0) | 0/27 (0) | 0/30 (0) | 0/26 (0) | 0/32 (0) | 0/34 (0) | 0/16 (0) | 0 (0) | 0/1 (0) | 0 (0) | 0 (0) | 0 (0) | 0/2 (0) | 0/1 (0) | 0/7 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (10) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 4 (8) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal sphincterotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 9 (10) | 0 (0) | 0 (0) | 3 (6) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT03482011/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03482011/SAP_001.pdf